CLINICAL TRIAL: NCT02448576
Title: A Phase III Randomized Controlled Trial of Prophylactic Cranial Irradiation in Patients With Advanced Triple Negative Breast Cancer Who Had a Response to First Line Chemotherapy
Brief Title: PCI in Advanced Triple Negative Breast Cancer Patients Who Response to 1st Line Chemotherapy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: wang shusen (Other)
Responsible Party: Sponsor-Investigator, wang shusen, Shusen Wang, M.D. Department of Medical Oncology, Sun Yat-sen University Cancer Center, Sun Yat-sen University
Organization: Sun Yat-sen University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: SYSU-5010-TNBC-PCI
Record Dates: First submitted 2015-05-05; First posted 2015-05-19 (Estimated); Last update posted 2017-06-01 (Actual); Status verified 2017-05

CONDITIONS: Breast Cancer; Brain Metastasis
Keywords: phase 3 randomized controlled trial; prophylactic cranial irradiation; triple negative breast cancer; brain metastasis; advanced breast cancer
MeSH Terms: conditions — Breast Neoplasms; Brain Neoplasms; Triple Negative Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PCI group (Experimental): Receiving prophylactic cranial irradiation after response to first line chemotherapy.
  Interventions: Radiation: prophylactic cranial irradiation
- observation group (No Intervention): Patients in the observation group do not receive prophylactic cranial irradiation after response to first line chemotherapy.

INTERVENTIONS:
Radiation: prophylactic cranial irradiation — Prophylactic cranial irradiation in patients with advanced triple negative breast cancer who had a response to first line chemotherapy
  Arms: PCI group

SUMMARY:
The purpose of this study is to compare whether prophylactic cranial irradiation in patients with advanced triple negative breast cancer who had a response to first line chemotherapy could prolong brain-metastasis free survival.

DETAILED DESCRIPTION:
This is a phase III, randomized, controlled, open, multicenter clinical trial, designed to assess the efficacy and safety of prophylactic cranial irradiation (PCI) in advanced triple negative breast cancer who response to the first line chemotherapy. Compare the PCI group with the observation group to evaluate brain metastasis-free survival,cumulative risk of brain metastases within 1 year,progression-free survival,overall survival,quality of life measured by the The Europe organization for research and treatment of cancer, Quality of life Questionnaire-cancer 30 (EORTC-QLQ-C30) questionnaire score and function of central nervous measured by the The Europe organization for research and treatment of cancer, Quality of life Questionnaire-brain cancer 20 (EORTC-QLQ-BN20) questionnaire score in women with advanced triple negative breast cancer who response to the first line chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent;
2. Age of 18 to 65 years;
3. Documented advanced breast cancer, clinical and pathological confirmed;
4. Immunohistochemical examination:ER<1%+, progestin receptor (PR)<1%+, HER-2 -/+ or HER-2(++)with negative result of FISH;
5. A response after four to eight cycles of first line chemotherapy;
6. Life expectancy longer than six months evaluated by investigator;
7. A performance status of 0 to 2, according to the criteria of the World Health Organization (with a higher score indicating a poorer performance status)
8. Less than grade 1( Common Terminology Criteria grade version 4.0) of treatment-related toxicities;
9. Adequate baseline organ function.

Exclusion Criteria:

1. History of another malignancy.
2. Pregnancy or gestation
3. Definite diagnosed of central nervous system (CNS)or leptomeningeal metastases
4. Serious cardiac illness or medical condition
5. Known history of related central nervous system or leptomeningeal disease
6. Cognition impairment or suffering from mental illness
7. Demand a long-term oral administration of psychotropic drugs
8. Have a concurrent disease or condition that may interfere with study participation, or any serious medical disorder that would interfere with the subject's safety (for example, active or uncontrolled infection, currently active/requiring anti-viral therapy hepatic or biliary disease)

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 326 (Estimated)
Dates: Start 2017-08 (Estimated); Primary Completion 2025-08 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
brain metastasis-free survival | eight years
  time from randomization to brain metastasis

SECONDARY OUTCOMES:
cumulative risk of brain metastases within 1 year | one year
  the percent of subjects occurring brain metastases with 1 year
progression-free survival | eight years
  time from randomization to disease progression or death(upon which happen earlier)
overall survival | eight years
  time from randomization to death
life quality score | eight years
  quality of life measured by the EORTC-QLQ-C30 questionnaire score
central nervous function score | eight years
  function of central nervous measured by the EORTC-QLQ-BN20 questionnaire score

CONTACTS AND LOCATIONS:
Overall Officials: Shusen Wang, Study Chair — Sun Yat-sen University
Locations (1):
- State Key Laboratory of Oncology in South China, Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

REFERENCES:
- [Background] Berghoff A, Bago-Horvath Z, De Vries C, Dubsky P, Pluschnig U, Rudas M, Rottenfusser A, Knauer M, Eiter H, Fitzal F, Dieckmann K, Mader RM, Gnant M, Zielinski CC, Steger GG, Preusser M, Bartsch R. Brain metastases free survival differs between breast cancer subtypes. Br J Cancer. 2012 Jan 31;106(3):440-6. doi: 10.1038/bjc.2011.597. Epub 2012 Jan 10. PMID 22233926
- [Background] Saip P, Cicin I, Eralp Y, Karagol H, Kucucuk S, Cosar Alas R, Yavuz E, Dincer M, Saglam E, Topuz E. Identification of patients who may benefit from the prophylactic cranial radiotherapy among breast cancer patients with brain metastasis. J Neurooncol. 2009 Jun;93(2):243-51. doi: 10.1007/s11060-008-9769-0. Epub 2008 Dec 20. PMID 19099196
- [Background] Le Scodan R, Jouanneau L, Massard C, Gutierrez M, Kirova Y, Cherel P, Gachet J, Labib A, Mouret-Fourme E. Brain metastases from breast cancer: prognostic significance of HER-2 overexpression, effect of trastuzumab and cause of death. BMC Cancer. 2011 Sep 19;11:395. doi: 10.1186/1471-2407-11-395. PMID 21929800
- [Background] Huang F, Alrefae M, Langleben A, Roberge D. Prophylactic cranial irradiation in advanced breast cancer: a case for caution. Int J Radiat Oncol Biol Phys. 2009 Mar 1;73(3):752-8. doi: 10.1016/j.ijrobp.2008.05.031. Epub 2008 Oct 26. PMID 18954943
- [Background] Tsukada Y, Fouad A, Pickren JW, Lane WW. Central nervous system metastasis from breast carcinoma. Autopsy study. Cancer. 1983 Dec 15;52(12):2349-54. doi: 10.1002/1097-0142(19831215)52:123.0.co;2-b. PMID 6640506
- [Background] Slotman B, Faivre-Finn C, Kramer G, Rankin E, Snee M, Hatton M, Postmus P, Collette L, Musat E, Senan S; EORTC Radiation Oncology Group and Lung Cancer Group. Prophylactic cranial irradiation in extensive small-cell lung cancer. N Engl J Med. 2007 Aug 16;357(7):664-72. doi: 10.1056/NEJMoa071780. PMID 17699816
- [Background] Auperin A, Arriagada R, Pignon JP, Le Pechoux C, Gregor A, Stephens RJ, Kristjansen PE, Johnson BE, Ueoka H, Wagner H, Aisner J. Prophylactic cranial irradiation for patients with small-cell lung cancer in complete remission. Prophylactic Cranial Irradiation Overview Collaborative Group. N Engl J Med. 1999 Aug 12;341(7):476-84. doi: 10.1056/NEJM199908123410703. PMID 10441603
- [Background] Ahn HK, Park YH, Lee SJ, Park S, Maeng CH, Park W, Choi DH, Hur SJ, Ahn JS, Im YH. Clinical implication of Time To Brain Metastasis (TTBM) according to breast cancer subtypes. Springerplus. 2013 Mar 28;2(1):136. doi: 10.1186/2193-1801-2-136. Print 2013 Dec. PMID 23667803
- [Background] Lin NU, Bellon JR, Winer EP. CNS metastases in breast cancer. J Clin Oncol. 2004 Sep 1;22(17):3608-17. doi: 10.1200/JCO.2004.01.175. PMID 15337811
- [Background] Bai B, Yuan ZY, Liu DG, Teng XY, Wang SS. Clinical features and survival analysis of different subtypes of patients with breast cancer brain metastases. Chin J Cancer. 2010 Apr;29(4):413-9. doi: 10.5732/cjc.009.10643. PMID 20346218
- [Background] Paterson AH, Agarwal M, Lees A, Hanson J, Szafran O. Brain metastases in breast cancer patients receiving adjuvant chemotherapy. Cancer. 1982 Feb 15;49(4):651-4. doi: 10.1002/1097-0142(19820215)49:43.0.co;2-x. PMID 7055779
- [Background] Carey LA, Ewend MG, Metzger R, Sawyer L, Dees EC, Sartor CI, Moore DT, Graham ML. Central nervous system metastases in women after multimodality therapy for high risk breast cancer. Breast Cancer Res Treat. 2004 Dec;88(3):273-80. doi: 10.1007/s10549-004-0999-3. PMID 15609130
- [Background] Al-Shamy G, Sawaya R. Management of brain metastases: the indispensable role of surgery. J Neurooncol. 2009 May;92(3):275-82. doi: 10.1007/s11060-009-9839-y. Epub 2009 Apr 9. PMID 19357955
- [Background] Fokstuen T, Wilking N, Rutqvist LE, Wolke J, Liedberg A, Signomklao T, Fernberg JO. Radiation therapy in the management of brain metastases from breast cancer. Breast Cancer Res Treat. 2000 Aug;62(3):211-6. doi: 10.1023/a:1006486423827. PMID 11072785
- [Background] Santarelli JG, Sarkissian V, Hou LC, Veeravagu A, Tse V. Molecular events of brain metastasis. Neurosurg Focus. 2007 Mar 15;22(3):E1. doi: 10.3171/foc.2007.22.3.2. PMID 17608351
- [Background] Gabos Z, Sinha R, Hanson J, Chauhan N, Hugh J, Mackey JR, Abdulkarim B. Prognostic significance of human epidermal growth factor receptor positivity for the development of brain metastasis after newly diagnosed breast cancer. J Clin Oncol. 2006 Dec 20;24(36):5658-63. doi: 10.1200/JCO.2006.07.0250. Epub 2006 Nov 13. PMID 17102066
- [Background] Tham YL, Sexton K, Kramer R, Hilsenbeck S, Elledge R. Primary breast cancer phenotypes associated with propensity for central nervous system metastases. Cancer. 2006 Aug 15;107(4):696-704. doi: 10.1002/cncr.22041. PMID 16826579